CLINICAL TRIAL: NCT04519151
Title: A Phase II, Open Lable, Single Arm, Trial to Determine Efficacy and Safety of Lenvatinib in Combination With Pembrolizumab for Platinum- Sensitive Recurrent Ovarian Cancer
Brief Title: Pembrolizumab and Lenvatinib for Platinum- Sensitive Recurrent Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Ronnie Shapira, M.D, Head onco-gynecological service, Principal Investigator, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7405-20
Record Dates: First submitted 2020-08-04; First posted 2020-08-19 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Neoplasm of Stomach; Ovarian Diseases; Genital Neoplasms, Female; Ovarian Epithelial Tumor; Urogenital Neoplasms; Neoplasms, Glandular and Epithelial
Keywords: Ovarian Cancer; Platinum sensitive; Ovarian Epithelial; Neoplasms; Genital Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Stomach Neoplasms; Ovarian Diseases; Genital Neoplasms, Female; Urogenital Neoplasms; Neoplasms, Glandular and Epithelial; Neoplasms | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Intervention Model Description: single arm
Masking Description: Open Lable
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lenvatinib 20 mg + Pembrolizumab 200 mg (Experimental): Participants will receive pembrolizumab 200 milligram (mg) administered by intravenous (IV) infusion on Day 1 of each 21-day cycle plus lenvatinib 20 mg administered orally (PO) once daily (QD) during each 21-day cycle for up to 35 cycles.
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg administered by IV infusion on Day 1 of each 21-day cycle.
  Other Names: KEYTRUDA®; MK-3475
Drug: Lenvatinib — 20 mg administered orally (PO) QD during each 21-day cycle.
  Other Names: LENVIMA®

SUMMARY:
This is a study of pembrolizumab (MK-3475, KEYTRUDA®) in combination with lenvatinib (E7080) for the treatment of platinum sensitive recurrent ovarian cancer. Participants will receive pembrolizumab and lenvatinib.

DETAILED DESCRIPTION:
This will be a phase-2, open-label, single-arm, single-center study to assess the effect of pembrolizumab and Lenvatinib combination therapy on platinum-sensitive recurrent ovarian cancer (ROC) patients.

Female patients 18 years of age or older with histologically-confirmed epithelial ovarian cancer (EOC) - excluding low grade tumors and mucinous histology - and documented disease recurrence following primary or interval debulking surgery and 1-2 prior lines of chemotherapy (including a frontline platinum-based regimen) and a platinum-free interval greater than 6 months will be eligible to enroll in the study.

Twenty-four patients will be included in the study. The study diagram is shown in Figure 1 and the schedule of assessments (SoA) is shown in Section 6.0. After signing the informed consent, eligible subjects according to the inclusion and exclusion criteria will receive oral Lenvatinib 20 mg once daily (QD) plus intravenous (IV) pembrolizumab 200 mg every three weeks (Q3W) until evident progressive disease by CT (RECIST), or unacceptable toxicity, or until completion of 35 treatment cycles with pembrolizumab.

Disease status will be evaluated radiologically by computed tomography (CT) every 9 weeks, in comparison to pretreatment CT, until progression. In case of study withdrawal due to other reasons, radiological evaluation will be maintained every 9 weeks until disease progression or patient's withdrawal of consent or a new anticancer regimen is given. Patients with contrast media allergy will undergo chest CT without contrast medium as well as abdominal and pelvic magnetic resonance imaging (MRI).

Toxicity will be graded by the National Cancer Institute Common Terminology Criteria for Adverse Events Ver. 5.0 (NCI-CTCAE). Dose reductions and modification of Lenvatinib will be performed according to the indications in Section 5.2.3. Pembrolizumab dose will not be reduced but the dose can be delayed for up to 9 weeks in case of toxicity which requires steroid.

treatment and steroids withdrawal (refer to Section 5.2.2 on pembrolizumab dose interruptions). Refer to section 5.2.4 for dose modifications for overlapping toxicities.

Health-related quality of life will also be evaluated. Collateral research will focus on potential biomarkers of response to treatment and on micro- and macro-environmental changes occurring during the course of treatment. To that end, tumor biopsies, stool and vaginal swabs and blood (plasma, serum and peripheral blood mononuclear cells (PBMC)) samples will be collected at Screening and during the study. Analyses will be performed to determine pre- and post-treatment changes as well as differences between responders to treatment and non-responders.

Participants who stop study treatment after receiving 35 administrations of pembrolizumab for reasons other than disease progression or intolerability, or participants who attain a complete response (CR) and stop study treatment may be eligible for up to 1 year of treatment with pembrolizumab (17 cycles) ± Lenvatinib upon experiencing disease progression (Second Course Phase). Participants who complete treatment with pembrolizumab after 35 cycles (approximately 2 years) or CR will continue to receive Lenvatinib alone until disease progression, development of unacceptable toxicity, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants who are at least 18 years of age on the day of signing informed consent, with histologically-confirmed diagnosis of EOC (except from low grade tumors and mucinous histology).
2. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow the contraceptive during the treatment period and for at least 120 days after the last dose of study treatment.
3. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
4. Have measurable disease at baseline based on RECIST 1.1. Lesions
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
6. Have received a front-line platinum-based regimen per local standard of care or treatment guideline following the primary or interval debunking surgery with radiologically documented disease recurrence no earlier than 6 months following completion of platinum-based therapy.

Note: Maintenance treatment following front-line treatment is permitted and counted together as part of the front-line treatment. Recurrence is evaluated since last platinum-based chemotherapy administration (for patients treated with maintenance bevacizumab or PARP inhibitors) Note: Patients that received maintenance immune checkpoint inhibitors will be eligible if progression was documented over 6 months since completion of the immunotherapy maintenance treatment.

Have received 0 to 1 line of chemotherapy for ROC (or 1 to 2 total prior lines counting the front line) and must have a PFI (or treatment-free interval) of >6 months for each treatment line.

8. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated.

9. Have adequately controlled blood pressure (BP) with or without antihypertensive medications 10. Have adequate organ function as defined by blood tests.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test
2. The participant is pregnant or breastfeeding at Screening or Baseline, or is expecting to conceive within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
3. The participant has received prior therapy with an anti-PD-1, anti-PD-L1 oranti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137) in the last 6 months (6 months are calculated from the last dose until study initiation).
4. The participant has received prior systemic anti-cancer therapy mAb, chemotherapy or targeted small molecule therapy within 4 weeks prior to the planned first dose of the study, including investigational agents within 4 weeks. For tyrosine kinase inhibitors (TKIs), other than lenvatinib, and hormonal therapy a shorter interval of 5 half-lives is allowed between prior therapy and study treatment initiation.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.
5. The participant has received prior lenvatinib.
6. The participant has received prior radiotherapy within 2 weeks of start of study treatment.
7. The patient had prior grade 3 immune related toxicity due to immune checkpoint inhibitors or non-infectious pneumonitis.
8. The participant has received more than 2 prior chemotherapy lines.
9. The participant has a history of tumor bleeding one month before study enrollment.
10. The participant has received a live vaccine within 30 days prior to the first dose of study drug.
11. The participant is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.

    Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
12. The participant has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.

    Note: The use of physiologic doses of corticosteroids is allowed.
13. The participant has a known active second/additional malignancy that is progressing or has required active treatment within the past 5 years Note: Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, in situ cervical cancer.
14. The participant has a known active CNS metastases and/or carcinomatous meningitis.

    Note: Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
15. The participant has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of excipients.
16. The participant has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

    Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
17. The participant has an active infection requiring systemic therapy.
18. The participant has a known history of human immunodeficiency virus (HIV 1/2 antibodies).
19. The participant has a known history of hepatitis B or known active hepatitis C virus
20. The participant has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
21. The participant has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
22. The participant has had an active allogenic tissue/solid organ transplant.
23. The participant has uncontrolled blood pressure
24. The participant has clinically significant electrolyte abnormalities that have not been corrected.
25. The participant has significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or cerebrovascular accident (CVA) within 6 months of the first dose of study drug, or cardiac arrhythmia associated with hemodynamic instability requiring medical treatment at Screening.
26. The participant has bleeding or thrombotic disorders, radiographic evidence of major blood vessel invasion/infiltration, or is at risk for severe hemorrhage.

    Note: The degree of tumor invasion/infiltration of major blood vessels (e.g. carotid artery) should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.
27. The participant has >1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours.
28. Prolongation of QTc interval to >480 ms.
29. Left ventricular ejection fraction (LVEF) below the institutional normal range as determined by multigated acquisition scan (MUGA) or echocardiogram (ECHO).
30. The participant has gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib.
31. The participant has a pre-existing Grade ≥3 gastrointestinal or non-gastrointestinal fistula.
32. The participant has a known intolerance to the study treatment (or any of its excipients).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
PFS of patients treated with pembrolizumab in combination with lenvatinib. | Up to approximately 27 months
  defined as the time from study treatment initiation to the first documented disease progression according to RECIST 1.1 or death from any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) in patients treated with a combination of pembrolizumab and lenvatinib. | Up to approximately 27 months
  defined as the percentage of evaluable patients with complete response (CR) or partial response (PR). Response will be evaluated by the Investigator according to RECIST 1.1.
Time to subsequent therapy (in months)- time from enrollment to next line of therapy initiation | Up to approximately 27 months
  defined as the time (in months) from initiation of treatment with pembrolizumab and Lenvatinib to subsequent chemotherapy treatment initiation.
Overall survival (OS) of the study population. | Up to approximately 27 months
  defined as the time from study treatment initiation to death due to any cause.
Impact of the treatment protocol on health-related quality of life using the QOL questionnaire (EORTC) QLQ-C30 | will be assessed at the pre-treatment visit and at the time of Tumor Imaging (schedualed or unschedualed with a ±3 day window. Additional assessment will be performed and at the end of treatment/discontinuation visit.
  To evaluate the impact of the treatment protocol on health-related quality of life (HR-QoL) as assessed by using the global score of the European Organization for the Research and Treatment of Cancer (EORTC) QLQ-C30.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Incidence of treatment-related adverse, serious adverse events, immune-related AEs | Up to approximately 27 months
  Safety and tolerability assessed by CTCAE v5.0.
Incidence of dose reductions | Up to approximately 27 months
  Safety and tolerability assessed by CTCAE v5.0.
The proportion of treatment discontinuation events related to the treatment combination | Up to approximately 27 months
  Safety and tolerability assessed by CTCAE v5.0.
Impact of the treatment protocol on health-related quality of life using the QOL questionnaire (EORTC) QLQ-OV28. | will be assessed at the pre-treatment visit and at the time of Tumor Imaging (schedualed or unschedualed with a ±3 day window. Additional assessment will be performed and at the end of treatment/discontinuation visit.
  To evaluate the impact of the treatment protocol on health-related quality of life (HR-QoL) as assessed by using the ovarian cancer-specific protocol, (EORTC) QLQ-OV28 for participants treated with Lenvatinib in combination with pembrolizumab.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

CONTACTS AND LOCATIONS:
Overall Officials: Ronnie Shapira, MD, Principal Investigator — Ronnie.Shapira@sheba.health.gov.il
Locations (1):
- Sheba Medical center, Ramat Gan, Israel